CLINICAL TRIAL: NCT02890394
Title: Effectiveness of the Suboccipital Inhibition Technique in Patients With Mechanical Neck Pain: a Pilot Study
Brief Title: Effectiveness of the Suboccipital Inhibition Technique in Patients With Mechanical Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alejandro Sánchez Tejada, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UAH
Record Dates: First submitted 2016-08-11; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Neck Pain; Myofascial Pain
Keywords: Neck Pain; Suboccipital inhibition; Physical Therapy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 minutes Group (Experimental): The group was perform the technique inhibition suboccipital two minutes, collecting data by measuring with algometer and test repositioning of the head before and after the technique.
  Interventions: Other: Suboccipital inhibition technique
- 4 minutes Group (Experimental): The group was perform the technique inhibition suboccipital four minutes, collecting data by measuring with algometer and test repositioning of the head before and after the technique.
  Interventions: Other: Suboccipital inhibition technique
- 8 minutes Group (Experimental): The group was perform the technique inhibition suboccipital eight minutes, collecting data by measuring with algometer and test repositioning of the head before and after the technique.
  Interventions: Other: Suboccipital inhibition technique
- not intervention Group (No Intervention): The not intervention group will be asked to lie supine on the table for ten minutes, collecting data by measuring with algometer and test repositioning of the head before and after laying.

INTERVENTIONS:
Other: Suboccipital inhibition technique — Suboccipital inhibition technique involves the placement of the hands of the physiotherapist under the patient's head so that fingers can feel the spinous processes of the cervical vertebrae. Then fingers slowly leads upward to contact the occipital condyles. At this point the investigator should gently move your fingers down, finding the space between the condyles and the spinous process of the axis. Remember that the atlas has no spinous process. Then, flexing the metacarpophalangeal joints at 90 degrees, slowly raises the skull
  Arms: 2 minutes Group; 4 minutes Group; 8 minutes Group

SUMMARY:
The project is based on checking the effectiveness of the technique of suboccipital inhibition in patients with mechanical neck pain. Suboccipital inhibition technique involves the placement of the hands of the physiotherapist under the patient's head so that fingers can feel the spinous processes of the cervical vertebrae. Then the fingers slowly leads upward to contact the occipital condyles. At this point the investigator should gently move your fingers down, finding the space between the condyles and the spinous process of the axis. Then, flexing the metacarpophalangeal joints at 90 degrees, slowly raises the skull. In this technique the investigator would be carrying out the relaxation of the suboccipital muscles: lower rectus capitis posterior, superior oblique head straight back and head higher. It is a technique used very often but without knowledge about the time needed for implementation. In several studies that have used the technique it has been maintained for 2.4 or 10 minutes without agreeing how long is necessary. The study will consist of three groups formed by patients with mechanical neck pain that they applied the technique two, four or ten minutes and a control group of patients with mechanical neck pain. The four groups were measured before and after treatment the pain threshold to pressure by algometer and conduct the test repositioning of the head to show any changes after application of the technique.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of full age .
2. ≥ 15/50 rating in the Neck Disability Index
3. Participants with good adhesion to the study .
4. Participants who have signed informed after appropriate informed consent.

Exclusion Criteria:

1. Cancer , inflammatory , infectious , vascular , neurological and metabolic processes.
2. Patients who are under medical treatment.
3. Patients with psychiatric illnesses.
4. Women : pregnancy.
5. Patients who have not signed the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change from pain threshold pressure after ten minutes from the suboccipital inhibition | It is measured at the beginning of the study. After ten minutes from the suboccipital inhibition is remeasured
  Three measurements were performed with a rest period of 30 seconds between each measurement.
Change from repositioning of the head after ten minutes from the suboccipital inhibition | It is measured at the beginning of the study. After ten minutes from the suboccipital inhibition is remeasured
  a target is placed on the wall in front of the subject at a distance of 90 cm and adjusted to align with the reference position of the head. a helmet with a laser on top is used. For each test subjects will be instructed to memorize the initial reference position by carrying out a maximum cervical rotation and returning to the reference position without speed limit. Subjects undertake 10 trials. Before each test, the examiner manually reposition the subject's head to the reference position. Once the subject is instructed to conduct the test measurement.

IPD SHARING:
Plan to Share IPD: No